CLINICAL TRIAL: NCT00486629
Title: Impact of a Community-based Obesity and Diabetes Prevention Program on Pregnant Outcomes in Pregnant Women
Brief Title: Impact of Diet and Exercise Activity on Pregnancy Outcomes
Acronym: IDEA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: The Lawson Foundation (Other); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Garry Shen, Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRT 2006-021
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Gestational Diabetes; Type 2 Diabetes
Keywords: Exercise; Diet; Pregnancy; Obesity; Macrosomia
MeSH Terms: conditions — Obesity; Diabetes, Gestational; Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Lifestyle questionnaire on mothers and offspring. Tests on glucose tolerance and epigenetic analysis in offspring.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Lifestyle intervention
  Interventions: Behavioral: Exercise and dietary education
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Exercise and dietary education — Exercise and dietary education. Aerobic exercise or walk for 3-5 times/day for 30-45 min/time from 20 weeks to 36 weeks of pregnancy. Dietary education on nutrition for healthy pregnancy through weekly class during pregnancy.
  Arms: Intervention

SUMMARY:
The general goal of the present study is to assess the impact of a community-based exercise and dietary intervention in pregnant women living in urban areas during and after their pregnancy on the reduction of the risks of both diabetes and obesity in mothers and their offspring.

We hypothesize that a community-based lifestyle intervention program during and after gestation may improve pregnancy outcomes in terms of reducing the risk of developing obesity or type 2 DM in mothers and their children.

DETAILED DESCRIPTION:
Impact of lifestyle intervention on excessive gestational weight gain

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy < 20 weeks.
* Expressed interest in study and willingness to consent to participate in the study.

Exclusion Criteria:

* Obstetric or medical contraindications for exercise according to 2002 SOCG guideline (ruptured membranes, preterm labor, incompetent cervix, hypertensive disorders of pregnancy, growth restricted fetus, placenta previa, persistent bleeding in 2nd or 3rd trimester, significant metabolic, cardiovascular, respiratory or systemic disorder) (5, 6).
* Pre-existing diabetes (except a history of GDM, but not in current pregnancy).
* Multiple gestations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2004-07; Primary Completion 2027-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Excessive weight gain during pregnancy | 2007-2023

SECONDARY OUTCOMES:
macrosomia, requirement of delivery procedures | 2007-2025

CONTACTS AND LOCATIONS:
Overall Officials: Garry Shen, MD PhD, Study Chair — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
1. Hui A, Back L, Ludwig S, Sellers E, McGavock J, Morris M, Bruce S, Shen GX. Lifestyle intervention on diet and exercise reduced excessive gestational weight gain in pregnant women under a randomized controlled trial. Br J Obstetr Gynecol 2012;119:70-77
  2. Hui AL, Back L, Ludwig S, Gardiner P, Sevenhuysen G, Dean HJ, Sellers E, McGavock J, Morris M, Jiang D, Shen GX. Effects of lifestyle intervention on dietary intake, physical activity level, and gestational weight gain in pregnant women with different pre-pregnancy Body Mass Index in a randomized control trial. BMC Pregnancy Childbirth. 2014;14:331. PMID:25248797

REFERENCES:
- [Result] Hui AL, Back L, Ludwig S, Gardiner P, Sevenhuysen G, Dean HJ, Sellers E, McGavock J, Morris M, Jiang D, Shen GX. Effects of lifestyle intervention on dietary intake, physical activity level, and gestational weight gain in pregnant women with different pre-pregnancy Body Mass Index in a randomized control trial. BMC Pregnancy Childbirth. 2014 Sep 24;14:331. doi: 10.1186/1471-2393-14-331. PMID 25248797
- [Result] Hui A, Back L, Ludwig S, Gardiner P, Sevenhuysen G, Dean H, Sellers E, McGavock J, Morris M, Bruce S, Murray R, Shen GX. Lifestyle intervention on diet and exercise reduced excessive gestational weight gain in pregnant women under a randomised controlled trial. BJOG. 2012 Jan;119(1):70-7. doi: 10.1111/j.1471-0528.2011.03184.x. Epub 2011 Oct 21. PMID 22017967